CLINICAL TRIAL: NCT05398666
Title: Investigation of Light Therapy in the Treatment Of Pain Caused By Osteoarthritis Of The Knee: A One-way Crossover Trial
Brief Title: Analgesic Potential of Light Therapy in Knee Osteoarthritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 154679
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Intervention Model Description: Patients will first receive White LED exposure, then they will be crossed over to Green LED exposure.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- White LED (Sham Comparator): Participants will be asked to use white LEDs for 1-2 hours/day in a dark room in their home.
  Interventions: Device: White LED light; Device: Green LED light
- Green LED (Experimental): Participants will be asked to use green LEDs for 1-2 hours/day in a dark room in their home.
  Interventions: Device: White LED light; Device: Green LED light

INTERVENTIONS:
Device: White LED light — Participants will be exposed to white LED lights (4 lux) in a dark room for 1-2 hours per day for 10 weeks.
Device: Green LED light — Participants will be exposed to green LED lights (4 lux) in a dark room for 1-2 hours per day for 10 weeks.

SUMMARY:
Managing joint pain is one of the main goals for treating osteoarthritis (OA) and other musculoskeletal disorders. Alleviating chronic pain pharmacologically has several potential drawbacks including diminishing efficacy, toxicity, adverse side-effects, and patient anxiety. Non-pharmacological approaches (eg. weight loss) have also been found to be effective at controlling joint pain and can provide supplementary benefits. The development of efficacious, alternative treatments for arthritis pain which provide analgesia without adverse side-effects would be advantageous.

Recently, preclinical and clinical studies have demonstrated that green ambient light using light-emitting diodes (LEDs) produced profound analgesia in animal models and chronic pain patients. Both migraineurs and fibromyalgia patients have both reported significant reductions in pain following 10 weeks of green LED exposure.

The investigators aim to assess the analgesic potential of green light therapy for people living with knee osteoarthritis. Participants will be asked to keep a pain diary for 4 weeks prior to light intervention. All participants will first use a white LED (20 lux) for 1-2 hours per day in a dark room at home for 10 weeks. Following a 2-week washout period without light use, participants will use a green LED (20 lux) for 1-2 hours per day in a dark room at home for 10 weeks. Following completion of the intervention, the investigator will assess changes in reported pain and quality of life. The investigators hypothesize that participants will have improvements in pain intensity and quality of life following treatment with green LEDs.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a progressive joint disease that affects 13% of Canadians. Managing joint pain is one of the main goals for treating OA and other musculoskeletal disorders. Alleviating chronic pain pharmacologically has several potential drawbacks including diminishing efficacy, toxicity, adverse side-effects, and patient anxiety. Current treatments consist mainly of oral nonsteroidal anti-inflammatories which are associated with significant side-effects such as higher risk of gastrointestinal (GI)ulcers and upper GI bleeds. Opioids as well are used but again present the risk that are associated with sedation, constipation and for some individuals substance disorders and addiction. Non-pharmacological treatments for OA pain may be beneficial.

Recently, preclinical and clinical studies have demonstrated that green ambient light using light-emitting diodes (LEDs) produced profound analgesia in chronic pain patients. Migraineurs exposed to this green light therapy (GLT) for 1-2 hours per day for 10 weeks reported a significant reduction in both headache days as well as headache intensity. Similarly, fibromyalgia patients treated with the same conditions reported a significant reduction in average pain intensity. Both patient groups also reported improvements in quality-of-life following treatment as measured by the EQ-5D-5L survey and, importantly, no adverse events were reported. White LEDs were used as a control in both trials and did not provide any analgesic benefit.

In pre-clinical rodent models, activation of the endogenous opioid system appears to be contributing to the analgesic effects of green light therapy. It is unknown if green light therapy may also be beneficial for osteoarthritis pain.

This study is a one-way crossover clinical design to determine whether exposure to green light therapy will improve pain in patients with knee osteoarthritis.

Initially, patients will receive White LED exposure (intensity: 4 lux, 1-2 hr/day), then they will be crossed over to Green LED exposure (wavelength 525nm, intensity: 4 lux, 1-2 hrs/day). The patients will not be told which one is the treatment and which one is the control.

Fourty patients attending the Chronic Pain Management Clinic with knee OA (as defined by the American College of Rheumatology guidelines) will be recruited to the study. Participants will be required to attend 4 visits during the 26 week study. In this study two light treatments will be tested (white LED vs green LED). Following the first clinic visit, we will ask participants to gather baseline pain information for 4 weeks without any light intervention (NRS-PI Pain Scale recorded in a pain diary). During weeks 5-15 participants will be exposed to white LEDs for 1-2 hours per day in a dark room at home, patients will then undergo a 2 week washout period without LED use. Green LEDs will be provided for home use for 1-2 hours per day (in a dark room) for the final 10 weeks. Visits to the clinic will follow the completion of both the white-light and green light treatments. Participants will be required to complete the NRS-PI Pain Scale every day and questionnaires at every visit. Questionnaires include the Brief Pain Inventory Short Form, The Western Ontario and McMaster Universities Arthritis Index (WOMAC), and the EuropQol EQ-5D-5L.

ELIGIBILITY:
Inclusion Criteria:

-Osteoarthritis of the knee according to American College of Rheumatology criteria: Knee pain with 3 of the following: age >50 years, stiffness less than 30 min, crepitus, bony tenderness, bony enlargement, no palpable warmth

* Moderate to severe pain, as defined by an average 7-day pain score of greater than 4.0 on an 11-point numerical rating scale for pain intensity (NRS-PI).
* All concurrent medications taken for any reason stable for 14 days
* Ability to follow protocol with reference to cognitive and situational factors (e.g. stable housing, ability to attend visits)
* Ability to read and write English
* Willing and able to give informed consent

Exclusion Criteria:

* Currently enrolled in other clinical trial involving a pharmaceutical treatment
* Arthroscopic surgery scheduled within 8 months of study initiation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain Score Diary | 24 weeks
  Change in mean daily pain diary score from baseline (average pain score over 7 days pre-treatment) to post treatment

SECONDARY OUTCOMES:
Western Ontario and McMaster University Arthritis Index (WOMAC) | 24 weeks
  Change in WOMAC score from baseline to post treatment
Global impression of change and satisfaction | 24 weeks
  Using the Global impression of change and satisfaction survey, changes in quality of life will be assessed following treatment
Brief Pain Inventory Short Form | 24 weeks
  Changes in reported pain will be assessed by comparing baseline and post-treatment responses

CONTACTS AND LOCATIONS:
Overall Officials: Karim Mukhida, MD, PhD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- NS Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No